CLINICAL TRIAL: NCT00408707
Title: Local Infiltration Analgesia With Ropivacaine Versus Placebo in Bilateral Knee Arthroplasty: a Placebo Controlled, Randomized, Double-Blinded Study.
Brief Title: Local Infiltration Analgesia With Ropivacaine Versus Placebo in Bilateral Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KF01320120
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Postoperative Pain
Keywords: local infiltration analgesia; postoperative pain; ropivacaine
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Procedure: local infiltration analgesia

SUMMARY:
The purpose of this study is to examine whether local infiltration analgesia (LIA) with Ropivacaine and adrenaline is effective in the treatment of postoperative pain after total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is increasingly common in the treatment of osteoarthrosis. Despite aggressive analgesic regimes, TKA is associated with moderate to severe postoperative pain, delaying mobilization and hospital discharge. A relatively new method for controlling postoperative pain after TKA is local infiltration analgesia (LIA) which consists of local infiltration with Ropivacaine and adrenaline.3 studies haved showed promising results of LIA, but none have documented a superior analgesic effect versus placebo.Patients receiving bilateral knee arthroplasty are recruited to receive LIA and placebo infiltration.The aim of the study is to demonstrate an analgesic effect of LIA versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for total knee arthroplasty
* must speak and understand Danish
* must be able to give oral and written consent

Exclusion Criteria:

* Alcohol or medicine abuse
* Treatment with opioids
* Allergy to local anaesthetics
* Severe obesity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain

SECONDARY OUTCOMES:
analgésia consumption
time to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Andersen, M.D., Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Andersen LO, Husted H, Otte KS, Kristensen BB, Kehlet H. High-volume infiltration analgesia in total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2008 Nov;52(10):1331-5. doi: 10.1111/j.1399-6576.2008.01777.x. PMID 19025523